CLINICAL TRIAL: NCT02939976
Title: Study of Access Site for Enhancing PCI in STEMI for Seniors (SAFE STEMI for Seniors)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for this study has been discontinued.
Sponsor: David Kong, M.D. (Other)
Collaborators: Medtronic Vascular (Industry); Volcano Corporation (Industry); Terumo Medical Corporation (Industry)
Responsible Party: Sponsor-Investigator, David Kong, M.D., Study Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00076262
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction
Keywords: ST-Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Single Vessel Disease (Active Comparator): Standard of care comparator for those subjects with single vessel coronary artery disease. Revascularization with Medtronic Resolute family of stents in infarct related artery; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device
  Interventions: Device: Single Vessel Disease; Device: Medtronic Resolute family of stents; Device: Terumo Glidesheath Slender; Device: Terumo TR Band Radial Compression Device
- Multi-vessel Disease, Culprit Vessel Only (Experimental): Subjects randomized to revascularization of infarct related artery only. Revascularization with Medtronic Resolute family of stents in infarct related artery; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device
  Interventions: Procedure: Multi-vessel Disease, Culprit Vessel Only; Device: Medtronic Resolute family of stents; Device: Terumo Glidesheath Slender; Device: Terumo TR Band Radial Compression Device
- Multi-vessel Disease, Complete Revascularization (Experimental): Subjects randomized to complete revascularization. Complete revascularization of all diseased arteries with Medtronic Resolute family of stents; Use of Volcano based pressure wires Verrata, Verrata Plus and any subsequent marketed Volcano pressure wire technology to determine which arteries to stent; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device
  Interventions: Procedure: Multi-vessel Disease, Complete Revascularization; Device: Medtronic Resolute family of stents; Device: Volcano based pressure wires Verrata, Verrata Plus and any subsequent marketed Volcano pressure wire technology; Device: Terumo Glidesheath Slender; Device: Terumo TR Band Radial Compression Device

INTERVENTIONS:
Device: Single Vessel Disease — Revascularization with Medtronic Resolute family of stents in infarct related artery; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device
  Arms: Single Vessel Disease
Procedure: Multi-vessel Disease, Culprit Vessel Only — Revascularization with Medtronic Resolute family of stents in infarct related artery; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device
  Arms: Multi-vessel Disease, Culprit Vessel Only
Procedure: Multi-vessel Disease, Complete Revascularization — Complete revascularization of all diseased arteries
  Arms: Multi-vessel Disease, Complete Revascularization
Device: Medtronic Resolute family of stents — Revascularization with Medtronic Resolute family of stents in infarct related artery
Device: Volcano based pressure wires Verrata, Verrata Plus and any subsequent marketed Volcano pressure wire technology — Complete revascularization of all diseased arteries
  Arms: Multi-vessel Disease, Complete Revascularization
Device: Terumo Glidesheath Slender — Possible use of Terumo Glidesheath Slender
Device: Terumo TR Band Radial Compression Device — Possible use of Terumo TR Band Radial Compression Device

SUMMARY:
Patients with partially blocked blood vessel(s) in their heart may need a medical procedure called "Percutaneous Coronary Intervention (PCI)" to open the narrowed blood vessel(s). The purpose of this study is to simultaneously address four potential advances in ST-Elevation Myocardial Infarction (STEMI) care for patients at least 65 years old. The investigators are looking to see if these advances can improve the outcome for these patients.

1. Opening the arteries with a Medtronic stent
2. Radial access (from wrist) success with a Medtronic stent
3. Checking the percent of blockage in the diseased artery/arteries using Volcano guide wires.
4. Reduced bleeding and vascular complications with radial arterial access for primary PCI in STEMI.

DETAILED DESCRIPTION:
Multicenter, randomized, open-label, unblinded, active and historical-controlled trial in which approximately 875 seniors undergoing urgent PCI from approximately 70 centers will be enrolled. All consented subjects will undergo attempted radial arterial access.

For DES (Drug Eluting Stent) eligible patients without randomization exclusion criteria and with multi-vessel disease identified during initial angiogram will be randomized by site in a ratio of 1:1 to IRA-only revascularization or iFR-guided complete revascularization. After randomization, subjects with stable TIMI-3 flow established in the IRA using the protocol specified treatment will proceed with the randomized procedure. Subjects in whom IRA reperfusion with TIMI-3 flow is not achieved will be treated according to clinical best practice standard of care independent of randomized procedure assignment and will not be considered protocol violations. These patients will be followed identically to all study patients.

After stent implantation, subjects will be contacted for follow-up at 30 days by the enrolling site and at 1 year by the DCRI Call Center.

Primary endpoint results will be reported after all subjects have completed 1 year (12 months) of clinical follow-up.

STEMI patients eligible for radial access:

* DES Eligible with single vessel Coronary Artery Disease (CAD) will receive DES to IRA
* DES Eligible with Multi-vessel CAD will randomize 1:1 to IRA-only revascularization or Instantaneous Wave Free Radio (iFR)-guided complete revascularization

ELIGIBILITY:
Inclusion Criteria

1. Have the capacity to understand and sign an informed consent or have a Legally Authorized Representative that can understand and sign an informed consent prior to initial arteriotomy access.
2. Age ≥ 60 years of age at the time of signing the informed consent and/or randomization.
3. Significant ST-elevation myocardial infarction or left bundle branch block (LBBB) on ECG with chest pain < 12 hours.
4. Accessible right or left radial artery conduit for PCI.
5. Physician intent to perform trans-radial PCI.
6. Willing to be contacted at 1 year by the DCRI Call Center

Study Randomization Inclusion Criteria

To be eligible for randomization in the 'IRA only vs. Complete Revascularization' phase of this trial, subjects must meet all of the above criteria and all of the following criteria subsequent to arterial access:

1. Subject eligible for DES implantation.
2. Angiographic multi-vessel CAD determined by local visual estimation.

Exclusion Criteria

1. Patient that have known medical conditions that would prevent or interrupt the recommended post procedure DES treatment regimen.
2. Patients that have known medical conditions that would prevent catheterization through the radial artery.
3. Patients that have known medical conditions that increase patient's risk above standard when using IFR.
4. Has had a cerebrovascular accident or transient ischemic neurological attack within the past 6 months.
5. Known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause noncompliance with the protocol.
6. Any condition associated with a life expectancy of less than 1 year.
7. Participation in another clinical study using an investigational agent or device within the past 3 months.

Study Randomization Exclusion Criteria If a subject who has been consented into the SAFE STEMI study develops or is found to have any of the following, they will not be eligible for randomization to an iFR guided complete revascularization vs. IRA-only primary PCI and will be excluded from the study.

1. Shock requiring pressors or mechanical circulatory assist support (IABP, Impella, ECMO, etc.) significant chronic renal disease (eGFR < 30) and/or on dialysis.
2. Other angiographic exclusions:

   * Single vessel CAD
   * Unprotected left main coronary artery disease
   * One or more major coronary distributions with CTO or indeterminate IRA
3. Clinical circumstances, which, in the judgment of the operator, preclude randomization.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Kong, MD, Principal Investigator — Duke University; Mitchell W Krucoff, MD, Study Chair — Duke University
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants with single vessel disease (SVD) were erroneously randomized and included in the intent-to-treat (ITT) population analyses.
Groups:
- Single Vessel Disease, Not Randomized: Standard of care comparator for those subjects with single vessel coronary artery disease who were not randomized.
  Revascularization with Medtronic Resolute family of stents in infarct related artery; Possible use of Terumo Glidesheath Slender and Terumo TR Band Radial Compression Device.
- Randomized to IRA Group: Participants randomly assigned to receive a coronary procedure involving evaluation by iFR to implant stents into multiple arteries (primary and others that are partially blocked).
  The Randomized to IRA group mainly includes participants with Multi-Vessel Disease, with the addition of two participants with single vessel disease (SVD) who were erroneously randomized to the IRA group and included in the intent-to-treat (ITT) population analyses.
- Randomized to iFR Group: Participants randomly assigned to receive a coronary procedure involving evaluation by iFR to implant stents into multiple arteries (primary and others that are partially blocked).
  The Randomized to iFR group mainly includes participants with Multi-Vessel Disease, with the addition of two participants with single vessel disease (SVD) who were erroneously randomized to the iFR group and included in the intent-to-treat (ITT) population analyses.
- Multi-vessel CAD, Non-randomized: Participants who had contraindications to performing the randomized procedure.
Period: Overall Study
Arm/Group | Single Vessel Disease, Not Randomized | Randomized to IRA Group | Randomized to iFR Group | Multi-vessel CAD, Non-randomized
Started | 177 | 82 | 77 | 91
Completed | 162 | 78 | 72 | 82
Not Completed | 15 | 4 | 5 | 9
Not completed — Lost to Follow-up | 7 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 4
Not completed — Due to early study closure | 4 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vessel Disease, Not Randomized | Randomized to IRA Group | Randomized to iFR Group | Multi-vessel CAD, Non-randomized | Total
Number analyzed (Participants) | 177 | 82 | 77 | 91 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.0) | 71.6 (7.4) | 72.0 (7.3) | 73.8 (7.7) | 71.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 25 | 18 | 26 | 123
  Male | 123 | 57 | 59 | 65 | 304
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 2 | 8 | 29
  Not Hispanic or Latino | 164 | 76 | 75 | 83 | 398
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 6 | 3 | 6 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 4 | 15
  White | 157 | 71 | 71 | 78 | 377
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 94 | 54 | 49 | 59 | 256
  Canada | 83 | 28 | 28 | 32 | 171

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated 1-year Infarct-related Artery Major Adverse Cardiac and Cerebrovascular Event (MACE)
Description: Defined as cardiac death, infarct artery target-vessel MI, or ischemia-driven index infarct related vessel revascularization (IIVR) by percutaneous or surgical methods.
Time Frame: 1 year
Population: Per SAP, all eligible enrolled participants who used Medtronic Drug Eluting stent during at least one CathPCI are included in this analysis. The rationale for the Metronic analysis population is that all subjects were intention-to-treat with a Resolute-family stent. So a study participant would have received the Medtronic stent for STEMI regardless of whether they were in the single-vessel, multivessel, or multivessel with FFR arm.
Measure: Count of Participants; unit: Participants
Groups:
- Medtronic Stent Population: Among all eligible enrolled participants, those who used Medtronic Drug Eluting stent during at least one CathPCI.
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 14

2. Primary Outcome: Adjudicated 1-year Modified CvLPRIT (Complete Versus Lesion-only Primary PCI Trial) MACE
Description: Defined as all-cause mortality, recurrent MI, heart failure (requiring hospitalization or 12 hour ER visit) or ischemia-driven revascularization for all treated arteries.
Time Frame: 1 year
Population: Per SAP, all eligible enrolled participants who were randomized are included. This includes 4 participants who were assigned to the Single-vessel CAD group and were subsequently randomized in error.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 9 | 5

3. Primary Outcome: Estimate of the Incidence Rate of Radial Artery Occlusion (RAO)
Description: Primary Observational Endpoint. Stratified by whether or not the Terumo TR Band was employed (use of the TR Band is recommended not required)
Time Frame: During procedure
Population: Per SAP, all eligible single vessel CAD (coronary artery disease) and multi-vessel subjects enrolled regardless of randomization in the study. Data were stratified by whether or not the Terumo TR Band was employed (use of the TR Band is recommended not required).
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Enrolled Population: All eligible single vessel CAD (coronary artery disease) and multi-vessel participants enrolled regardless of randomization in the study.
Arm/Group | Eligible Enrolled Population
Number analyzed (Participants) | 427
Participants
  TR Band: number analyzed (Participants) | 329
  TR Band | 0
  Without having TR Band: number analyzed (Participants) | 98
  Without having TR Band | 0

4. Primary Outcome: Estimate of the Incidence Rate of Radial Artery Occlusion (RAO)
Description: Primary Observational Endpoint - Stratified by whether or not the Terumo TR Band was employed (use of the TR Band is recommended not required)
Time Frame: 30 day
Population: Per SAP, data were stratified by whether or not the Terumo TR Band was employed (use of the TR Band is recommended not required)
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Enrolled Population
Number analyzed (Participants) | 427
Participants
  TR band: number analyzed (Participants) | 329
  TR band | 0
  Without having TR Band: number analyzed (Participants) | 98
  Without having TR Band | 0

5. Secondary Outcome: Adjudicated Death (All Causes)
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 14

6. Secondary Outcome: Adjudicated Death (All Causes)
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 2

7. Secondary Outcome: Adjudicated Cardiac Death
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 11

8. Secondary Outcome: Adjudicated Cardiac Death
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 0

9. Secondary Outcome: Adjudicated Nonfatal (re-) MI Myocardial (Infarction)
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 4

10. Secondary Outcome: Adjudicated Nonfatal (re-) MI
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 4

11. Secondary Outcome: Adjudicated Index Infarct Related Vessel (re-) MI
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 0

12. Secondary Outcome: Adjudicated Index Infarct Related Vessel (re-) MI
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 0

13. Secondary Outcome: Adjudicated Index Infarct Related Lesion Revascularization (IILR) (Ischemia Driven)
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 1

14. Secondary Outcome: Adjudicated Index Infarct Related Lesion Revascularization (IILR) (Ischemia Driven)
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 2

15. Secondary Outcome: Adjudicated Index Infarct Vessel Revascularization (IIVR) (Ischemia Driven)
Description: Efficacy endpoint
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 4

16. Secondary Outcome: Adjudicated Index Infarct Vessel Revascularization (IIVR) (Ischemia Driven)
Description: Efficacy endpoint
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 3

17. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite/Probable Stent Thrombosis
Description: Safety endpoint
Time Frame: Post-Procedure (0-24 hours post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 4

18. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite/Probable Stent Thrombosis
Description: Safety endpoint
Time Frame: 30 days (>24 hours through 30 days post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 4

19. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite/Probable Stent Thrombosis
Description: Safety endpoint
Time Frame: 1 year (>30 days post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 2

20. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite Stent Thrombosis
Description: Safety endpoint
Time Frame: Post-procedure (0-24hr post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 3

21. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite Stent Thrombosis
Description: Safety endpoint
Time Frame: 30 days (>24hr to 30 days post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 1

22. Secondary Outcome: Adjudicated Academic Research Consortium (ARC) Definite Stent Thrombosis
Description: Safety endpoint
Time Frame: 1 year (>30 days post stent)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 2

23. Secondary Outcome: Adjudicated Stroke
Time Frame: Post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 2

24. Secondary Outcome: Adjudicated Stroke
Time Frame: Baseline to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 0

25. Secondary Outcome: Adjudicated Stroke
Time Frame: Day 31 to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Stent Population
Number analyzed (Participants) | 362
Participants | 0

26. Secondary Outcome: Adjudicated Death (All Causes)
Time Frame: Baseline to 30 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 4 | 3

27. Secondary Outcome: Adjudicated Death (All Causes)
Time Frame: Day 31 to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 0 | 0

28. Secondary Outcome: Adjudicated Cardiac Death (All Causes)
Time Frame: Baseline to 30 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 3 | 3

29. Secondary Outcome: Adjudicated Cardiac Death (All Causes)
Time Frame: Day 31 to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 0 | 0

30. Secondary Outcome: Heart Failure (Requiring Hospitalization or 12 Hour ER Visit)
Time Frame: Baseline to 30 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 1 | 0

31. Secondary Outcome: Heart Failure (Requiring Hospitalization or 12 Hour ER Visit)
Time Frame: Day 31 to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 0 | 0

32. Secondary Outcome: Ischemia-driven Revascularization for Index Infarct Vessel Revascularization (IIVR) or Any Treated Index Non-infarct Related Vessels (INIVR)
Time Frame: 30 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 0 | 0

33. Secondary Outcome: Adjudicated Stroke
Time Frame: Baseline to 30 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 2 | 0

34. Secondary Outcome: Adjudicated Stroke
Time Frame: Day 31 to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
Participants | 0 | 0

35. Secondary Outcome: Incidence of RAO, Stratified by Whether or Not the Terumo TR Band Was Employed in Combination With GlideSheath Slender
Description: Secondary Observational Endpoint
Time Frame: 30 days
Population: Per SAP, all eligible enrolled participants who used Terumo products during at least one CathPCI. Terumo products include Terumo Glidesheath Slender and/or TR Band.
Measure: Number; unit: number of events
Groups:
- Terumo Population: All eligible enrolled participants who used Terumo products during at least one CathPCI. Terumo products include Terumo Glidesheath Slender and/or TR Band.
Arm/Group | Terumo Population
Number analyzed (Participants) | 329
number of events
  Without TR Band: number analyzed (Participants) | 34
  Without TR Band | 0
  On TR Band: number analyzed (Participants) | 295
  On TR Band | 0

36. Secondary Outcome: Site Reported Time to Achieve Hemostasis
Description: Secondary Observational Endpoint - Time to hemostasis stratified by whether the Terumo TR Band was employed
Time Frame: Post-procedure
Population: Enrolled participants who experienced hemostasis are included in the analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eligible Enrolled Population
Number analyzed (Participants) | 126
minutes
  Participants with Terumo TR Band: number analyzed (Participants) | 109
  Participants with Terumo TR Band | 249.44 (210.46)
  Participants without Terumo TR Band: number analyzed (Participants) | 17
  Participants without Terumo TR Band | 86.59 (56.79)

37. Secondary Outcome: Site Reported Time to Achieve Hemostasis
Description: Secondary Observational Endpoint - Time to hemostasis stratified by whether the Terumo TR Band was employed
Time Frame: Post-procedure
Population: Enrolled participants who experienced hemostasis are included in the analysis
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Eligible Enrolled Population
Number analyzed (Participants) | 126
minutes
  Participants with Terumo TR Band: number analyzed (Participants) | 109
  Participants with Terumo TR Band | 228 [94 to 350]
  Participants without Terumo TR Band: number analyzed (Participants) | 17
  Participants without Terumo TR Band | 96 [60 to 138]

38. Secondary Outcome: Incidence Rate of Cross Over From the Initial Access Point to Another Stratified by Whether or Not Terumo Slender GlideSheath Was Employed
Time Frame: During procedure
Population: Enrolled participants with non-missing GlideSheath status
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Enrolled Population
Number analyzed (Participants) | 421
Participants
  GlideSheath = No: number analyzed (Participants) | 86
  GlideSheath = No | 9
  GlideSheath = Yes: number analyzed (Participants) | 335
  GlideSheath = Yes | 16

39. Secondary Outcome: Incidence Rate of Access Success
Description: Access success is defined as successfully deploying the stent through the right or left radial artery stratified by whether or not Terumo Slender GlideSheath was employed
Time Frame: During procedure
Population: The outcome required several parameters from medical records to determine access success. However, these parameters were not collected before the study termination, therefore, this Outcome Measure was not collected.
Groups:
- Terumo Population: Per SAP, all eligible enrolled participants who used Terumo products during at least one CathPCI. Terumo products include Terumo Glidesheath Slender and/or TR Band.
Arm/Group | Terumo Population
Number analyzed (Participants) | 0

40. Other Pre Specified Outcome: Medtronic Resolute® Family of Stents - Site Determination of Procedure Success
Description: Site determination of procedure success, defined as lesion success without the occurrence of in-hospital death, nonfatal MI, stroke, or emergency Endpoints for Evaluating iFR Guided iFR-Guided Complete Revascularization in STEMI.
Time Frame: During index procedure in-hospitalization
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Medtronic Resolute® Family of Stents - Site Determination of Lesion Success
Description: Site determination of lesion success, defined as attainment of less than 20% residual stenosis using any percutaneous method at the time of the index procedure.
Time Frame: During index procedure
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Medtronic Resolute® Family of Stents - Site Determination of Device Success
Description: Site determination of device success, defined as attainment of less than 20% residual stenosis of the infarct related lesion at the time of the index procedure (IILR) using only the study stent.
Time Frame: During index procedure
Reporting Status: Not Posted

43. Other Pre Specified Outcome: iFR Guided Revascularization - Site Reported Index Hospitalization Bleeding and Vascular Complication Defined as Bleeding or Vascular Complication Requiring Intervention
Time Frame: During procedure
Reporting Status: Not Posted

44. Other Pre Specified Outcome: iFR Guided Revascularization With Volcano Based Pressure Wires Verrata®, Verrata Plus® and Any Subsequent Marketed Volcano Pressure Wire Technology - Total Procedure Time
Time Frame: During procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
minutes | 54.54 (24.39) | 65.91 (29.90)

45. Other Pre Specified Outcome: iFR Guided Revascularization With Volcano Based Pressure Wires Verrata®, Verrata Plus® and Any Subsequent Marketed Volcano Pressure Wire Technology - Total Contrast Used
Time Frame: During procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Randomized to IRA Group | Randomized to iFR Group
Number analyzed (Participants) | 82 | 77
mL | 144.5 (83.5) | 162.4 (72.3)

46. Other Pre Specified Outcome: Occurrence of Renal Insufficiency
Description: Device Performance Endpoint for evaluating iFR Guided iFR-Guided Complete Revascularization in STEMI. Renal insufficiency is defined as increase from baseline creatinine of at least 0.5 mg/dL or at least 25%
Time Frame: 48-72 hours post-procedure
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Occurrence of Renal Insufficiency
Description: as for outcome 46
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: SAEs and AEs were assessed up to 30 days. All-cause mortality is reported up to 1 year.
Arm/Group | Single Vessel Disease, Not Randomized | Randomized to IRA Group | Randomized to iFR Group | Multi-vessel CAD, Non-randomized
All-Cause Mortality (participants affected / at risk) | 10/177 | 4/82 | 3/77 | 6/91
Serious Adverse Events (participants affected / at risk) | 1/177 | 0/82 | 0/77 | 0/91
Other Adverse Events (participants affected / at risk) | 0/177 | 0/82 | 0/77 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Vessel Disease, Not Randomized (N=177) | Randomized to IRA Group (N=82) | Randomized to iFR Group (N=77) | Multi-vessel CAD, Non-randomized (N=91)
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02939976/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT02939976/SAP_001.pdf